CLINICAL TRIAL: NCT05840692
Title: The Effect of Anti Depressive Medicine on Adrenal Activity, Glucose Metabolism, Physical and Mental Health in Polycystic Ovary Syndrome. -A Randomised, Double Blinded, Placebo Controlled Study.
Brief Title: The Effect of Escitalopram in PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Andersen, Clinical professor, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: herbert4
Record Dates: First submitted 2013-05-30; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, doctors, alle people involved in analyses
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cipralex (Active Comparator): Escitalopram 20 mg x 1 for 12 weeks
  Interventions: Drug: Placebo
- Placebo (Placebo Comparator): Placebo 20 mg x 1 for 12 weeks
  Interventions: Drug: Escitalopram 20 mg

INTERVENTIONS:
Drug: Escitalopram 20 mg — Antidepressant
  Arms: Placebo
Drug: Placebo
  Arms: Cipralex

SUMMARY:
In a randomized study the investigators aim to characterize the effect of antidepressive medicine on quality of life, body composition, adrenal activity and glucose metabolism in PCOS.

PCOS is a common endocrine disorder characterized by adrenal and ovarian hyperandrogenaemia, anovulation and insulin resistance. The pathogenesis of PCOS may be described by a vicious cycle involving insulin resistance which stimulates ovarian and adrenal hyper androgenaemia and leads to abdominal obesity, causing increased risk for diabetes and cardiovascular disease. Adrenal hyperactivity is associated with depression. Antidepressive medicine may normalize pituitary-adrenal activity and in animal studies antidepressive medicine improved adrenal hyperactivity and normalized insulin sensitivity.

DETAILED DESCRIPTION:
Clinical study Effects of antidepressive treatment on quality of life, insulin sensitivity and cortisone metabolism in PCOS.

Hypothesis Participants with PCOS have increased hypothalamic-pituitary-adrenal activity compared to healthy women. Antidepressive treatment improves quality of life, cortisone and glucose turnover.

Design A randomized controlled study in 40 PCOS patients who are treated with cipralex or placebo for 12 weeks. Before and after the treatment period the patients have a physical examination, a whole body dexa scan and fasting blood samples. Hypothalamic-pituitary-adrenal is measured by 24 hour samples of cortisone metabolites, 60 minutes ACTH test with basal and stimulated measurement of cortisone and 17-hydroxyprogesterone. Glucose metabolism is examined by oral glucose tolerance test. Biopsies of muscle and fat are also performed.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25 and <5
* Age 18-45 years
* Two of the following 1: an/oligomenorhea, 2: Hirsutism or hyper androgenaemia, 3: PCO in trans vaginal ultrasound
* Other diagnoses excluded

Exclusion Criteria:

* Post menopausal
* Diabetes
* Eating disorder
* Psychiatric disorder
* Usage of oral anticonceptives or metformin
* Pregnancy or planned pregnancy in the treatment period
* Non-caucasian
* Epilepsy
* Allergy to the medicine

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Adrenal activity in urine | 12 weeks
  Cortisol in 24 h urine
Adrenal activity during stimulationtest | 12 weeks
  Cortisol during 60 min ACTH test

SECONDARY OUTCOMES:
Glucose assesment by 3 hour oral glucose tolerance test (OGTT) | 12 weeks
  Glucose
  - Muscle and fat biopsy

OTHER OUTCOMES:
Quality of life, SF36 | 12 weeks
  SF36
  - accelerometer i 7 days
Quality of life, VAS | 12 weeks
  VAS

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Andersen, DMSci, Principal Investigator — Odense University Hospital
Locations (1):
- Odense Universitetshospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided